CLINICAL TRIAL: NCT01443741
Title: Evaluation of Interests of the Functional Insulin Therapy (FIT Therapy) on Metabolic Control, Hypoglycemia Prevention and Life Quality of Diabetics Children Insulin-dependent Treated With Insulin Pump.
Brief Title: Evaluation of Interests of FIT Therapy on Diabetics Children Insulin-dependent
Acronym: DIABFIT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC 2009- 03
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Diabetes Insulin Dependent
Keywords: FIT Therapy; Diabetes mellitus; Insulin pump; Pediatric
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FIT Therapy (Active Comparator): Patient with functional insulin therapy
  Interventions: Other: Therapeutic education
- Traditional way (Active Comparator): Patient with traditional way
  Interventions: Other: Therapeutic education

INTERVENTIONS:
Other: Therapeutic education — Specific program for FIT Therapy and specific program for traditional way
  Other Names: Functional insulin therapy; Traditional way (fixed doses of insulin)

SUMMARY:
Evaluation of interests of the functional insulin therapy (FIT Therapy) on metabolic control, hypoglycemia prevention and life quality of diabetics children insulin-dependent treated with insulin pump.

DETAILED DESCRIPTION:
Open multicenter randomized study of one year, evaluating two groups of 44 children with diabetes mellitus (diabetes over 1 year) treated with insulin pump, one group by traditional way (fixed doses of insulin and meals providing stable quantities complex carbohydrates) and the other group by FIT Therapy.

ELIGIBILITY:
Inclusion Criteria:

* aged 1-17 years
* diabetic for at least 1 year
* whose HbA1c is between 7.6 and 10% (7.6% <HbA1C <10%)
* treated with insulin pump
* agreeing to perform at least three blood glucose/day
* willing to follow the treatment with functional insulin therapy if necessary

Exclusion Criteria:

* Ages <1 year or> 17 years
* Duration of diabetes <1 year
* HbA1c <7.6% or HbA1c> 10%
* Treatment-by multiple injections
* Mental disability
* Refusal to adhere to the constraints of the study
* Language barrier, preventing any understanding or cooperation
* Eating behavior-type anorexia or bulimia
* Pregnancy
* Use of alcohol or drugs
* Severe chronic or genetic pathology other than diabetes
* Participation in another clinical study or refusal to participate in the study

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Variation in HbA1c | One year
  Variation in HbA1c from baseline in the study (M0) and 1 year later the beginning of the program (M12) for assess the importance of the FIT Therapy to improve metabolic control of children with diabetes mellitus treated with subcutaneous insulin pump.

SECONDARY OUTCOMES:
Severe hypoglycemia over 6 months and quality of life | One year and six months
  Number of severe hypoglycemia over 6 months (M6 to M12 and evolution of quality of life assessed by validated questionnaries in children with diabetes (WHO questionnary items 5, 27 KIDSCREEN questionnary, DISABKID questionnary).

CONTACTS AND LOCATIONS:
Overall Officials: Régis Coutant, MD PhD, Principal Investigator — UH Angers
Locations (6):
- France (6):
  - University Hospital of Lyon, Lyon, Auvergne-Rhône-Alpes
  - University Hospital of Brest, Brest, Brittany Region
  - University Hospital of Tours, Tours, Centre-Val de Loire
  - University Hospital of Toulouse, Toulouse, Midi-Pyrénées
  - University Hospital of Angers Service of Pediatric Diabetology and Endocrinology, Angers, Pays de Loire
  - University Hospital of Nantes, Nantes, Pays de Loire

REFERENCES:
- [Background] Langewitz W, Wossmer B, Iseli J, Berger W. Psychological and metabolic improvement after an outpatient teaching program for functional intensified insulin therapy (FIT). Diabetes Res Clin Pract. 1997 Sep;37(3):157-64. doi: 10.1016/s0168-8227(97)00071-5. PMID 9306036
- [Background] Hartemann-Heurtier A, Sachon C, Masseboeuf N, Corset E, Grimaldi A. Functional intensified insulin therapy with short-acting insulin analog: effects on HbA1c and frequency of severe hypoglycemia. An observational cohort study. Diabetes Metab. 2003 Feb;29(1):53-7. doi: 10.1016/s1262-3636(07)70007-1. PMID 12629448
- [Background] Samann A, Muhlhauser I, Bender R, Kloos Ch, Muller UA. Glycaemic control and severe hypoglycaemia following training in flexible, intensive insulin therapy to enable dietary freedom in people with type 1 diabetes: a prospective implementation study. Diabetologia. 2005 Oct;48(10):1965-70. doi: 10.1007/s00125-005-1905-1. Epub 2005 Aug 18. PMID 16132954
- [Background] Lowe J, Linjawi S, Mensch M, James K, Attia J. Flexible eating and flexible insulin dosing in patients with diabetes: Results of an intensive self-management course. Diabetes Res Clin Pract. 2008 Jun;80(3):439-43. doi: 10.1016/j.diabres.2008.02.003. Epub 2008 Mar 18. PMID 18353485
- [Background] Grimm JJ, Ybarra J, Berne C, Muchnick S, Golay A. A new table for prevention of hypoglycaemia during physical activity in type 1 diabetic patients. Diabetes Metab. 2004 Nov;30(5):465-70. doi: 10.1016/s1262-3636(07)70144-1. PMID 15671916